CLINICAL TRIAL: NCT06356246
Title: Oral Health Status of Cystic Fibrosis Patients. An Online Survey in Collaboration With the Vaincre la Mucoviscidose Patient Association.
Acronym: E-MUCODENT
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Vaincre la Mucoviscidose (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240363
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cystic Fibrosis
Keywords: Oral quality of life; Periodontal disease; Oral health habits; Dental diseases
MeSH Terms: conditions — Cystic Fibrosis; Periodontal Diseases; Stomatognathic Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cystic Fibrosis (CF) is a rare hereditary disease with autosomal recessive transmission, affecting 1 in 4700 births in France. Numerous studies have explored the links between oral health and CF, predominantly focusing on a children population. These studies reveal hyposalivation, a risk of dental erosion, an increased prevalence of enamel structural defects, but a reduced prevalence of dental caries in CF children, potentially explained by better oral hygiene. Periodontal disease does not appear to be increased in this population, while the oral quality of life of CF patients has been insufficiently studied.

Today, emerging challenges arise due to the increased life expectancy of CF patients, attributed to the rise of modulators such as Kaftrio®, resulting in an adult-majority population in France. The study of periodontal diseases, associated with oral dysbiosis, becomes relevant as they represent bacterial reservoirs that could impact respiratory complications in CF patients.

To deepen understanding of the links between oral health and CF, as well as to improve oral health of these patients, it is crucial to update the specific oral profile of this population. A cross-sectional survey using a questionnaire is proposed to include a large number of CF patients in France, aiming for real-life data. This questionnaire is constructed around internationally recognized tools for comparative analysis with normative data. Collaboration with the Patients Association "Vaincre la Mucoviscidose" (VLM) facilitates questionnaire creation, dissemination, and interpretation of results.

DETAILED DESCRIPTION:
Cystic Fibrosis (CF) is a rare hereditary disease with autosomal recessive transmission, affecting 1 in 4700 births in France. It is characterized by a mutation in the CFTR gene (Cystic Fibrosis Transmembrane conductance Regulator), which codes for a channel regulating chloride ion transport on the surface of epithelial cells in exocrine glands. While its primary impact is pulmonary, various systemic effects, including oral manifestations, are documented.

Several studies have explored the links between oral health and CF. They reveal the existence of hyposalivation associated with an increased risk of dental erosion, an elevated prevalence of enamel structural defects, and a reduced incidence of dental caries in CF children. Studies on the relationship between periodontal disease (periodontitis) and CF have shown no significant difference between CF patients and the general population. The oral quality of life in CF patients, measured by the OHIP-14 (Oral Health Impact Profile), a 14-item questionnaire, is also of interest, with only one study to date assessing this dimension in a population of minors.

These studies, often limited in scope, primarily focus on a CF population consisting mainly of children and young adults. In recent years, improved CF management has increased the median lifespan, exceeding 50 years (maximum age recorded in 2022: 85 years). New challenges arise due to the growing adult CF population. Additionally, the oral cavity acts as a bacterial reservoir at the entrance of airways, impacting chronic pulmonary conditions such as Chronic Obstructive Pulmonary Disease (COPD). Bacteria found in the oral environment (e.g. P. aeruginosa) are also identified in CF patients' lungs. The study of oral bacterial diseases in CF patients is of particular interest.

Therefore, to enhance knowledge on the links between oral health and CF and improve dental care for CF patients, updating the specific dental profile of this population with specific needs is necessary.

Objective and Methods : The proposed research is a questionnaire-based health data study aiming to improve knowledge of the links between oral health and CF. Due to early CF diagnosis, improved patient care, and innovative therapies in recent years, the median lifespan of CF patients has increased. While the disease traditionally affected only children, the adult population became the majority in France, representing nearly 60% in 2020. Yet, there is limited data on the oral health status of these patients, despite the importance of oral health for overall health and patient quality of life. The questionnaire seeks to collect data on socio-professional categories, medical history, dental care, periodontal/tooth wear/caries risk, mouth dryness, and oral quality of life, to identify real-life oral care needs for CF patients. The questionnaire, developed in collaboration with the "Vaincre La Mucoviscidose" association, uses reference tools from international literature :

Periodontal Risk Screening Score Tooth Decay/Tooth Wear Risk Score Oral Quality of Life OHIP-14 Mouth Dryness Shortened version of Xerostomia Inventory

Additionally, the study aims to assess whether CF patients follow the recommendations of the French Union for Oral Health 2022 for check-ups (2/year for chronic diseases) and good oral hygiene practices (2 brushings of 2 minutes/day with a soft toothbrush, daily interdental brushing, and fluoridated toothpaste). This study encompasses all adult CF patients in France, numbering over 4000 (4577 adult CF patients according to the French CF registry data report 2022 .The research is based on a Lime Survey questionnaire that will be distributed to all cystic fibrosis patients in France, via the association's newsletter and the Vaincre La Mucoviscidose social networks, as well as posters in the waiting rooms of these patients' care centers (Filière MucoCFTR). The research is monocentric, carried out by Prof. Gosset in the oral medicine department of Hôpital Charles Foix AP-HP.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient (> 18 years old)
2. Cystic fibrosis patient
3. Patient who speaks and understands French well enough to read and understand the study information leaflet.
4. Patient does not object to participation in the study

Exclusion Criteria:

NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with cystic fibrosis treated in France
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Periodontal Risk Screening Score PESS | 3 months
  The Periodontal Screening Score (PESS) is a simple screening method based on 10 questions that helps identify individuals who may be at risk of periodontitis. It was developped and published by Carra et al in 2018.
  Score values: 0 up to 13, higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Assess the adherence to good oral hygiene practices and dental follow-up in adult CF patients according to French Union for Oral Health (UFSBD) 2021 | 3 months
  From the questionnaire: % of patients declaring to have a bi-annual follow-up and performing 2 brushing sessions of 2 min/day with a soft toothbrush, daily interdental brushing and fluoride toothpaste.
Evaluate the risk of dental caries and tooth wear | 3 months
  For the evaluation : use of the questions from the RestoData national cross-sectional clinical study "Evaluation of direct and indirect partial coronal dental fillings in a network of private clinical research and university hospital odontology departments", led by Prof. Grosgogeat, Hospices civils de Lyon.
Assess the oral quality of life | 3 months
  use of OHIP-1 Score values: 0 up to 7, higher scores mean a worse outcome.
Evaluate oral dryness | 3 months
  selected questions from the Xerostomia Inventory (shortened version). Score values: 5 up to 25, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Marjolaine GOSSET, Ivry-sur-Seine, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor.
Access Criteria: Researchers who provide a methodologically sound proposal.